CLINICAL TRIAL: NCT02180646
Title: Effect of a High Protein Breakfast on Glycemic Control, Insulin Sensitivity, and Beta Cell Function in Individuals With Type 2 Diabetes (T2D)
Brief Title: Impact of Breakfast Composition on Glycemic and Incretin Responses in Individuals With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: American Egg Board (Other)
Responsible Party: Principal Investigator, Jill Kanaley, professor, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: b2d2-01
Record Dates: First submitted 2014-06-30; First posted 2014-07-03 (Estimated); Results first posted 2017-01-18 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Type 2 Diabetes
Keywords: GLP-1; GIP; second meal phenomena; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Carb then High Protein Breakfast (Active Comparator): A high carbohydrate breakfast - 500 kcal (15% protein, 65% CHO, 20% fat) followed by a 7-day washout period, and then 7 days of eating a high protein breakfast - 500 kcal (35% protein, 45% CHO, 20% fat).
  Interventions: Other: High protein breakfast; Other: High carb breakfast
- High Protein then High Carb Breakfast (Active Comparator): A high protein breakfast - 500 kcal followed by a 7-day washout period, and then 7 days of eating a high carbohydrate breakfast - 500 kcal (35% protein, 45% CHO, 20% fat)
  Interventions: Other: High protein breakfast; Other: High carb breakfast

INTERVENTIONS:
Other: High protein breakfast — a high protein breakfast - 500 kcal (35% protein, 45% CHO, 20% fat)
Other: High carb breakfast — a high carbohydrate breakfast - 500 kcal (15% protein, 65% CHO, 20% fat)

SUMMARY:
This study examined the effect of a high protein or high carbohydrate breakfast on the glucose and insulin response following the breakfast meal, as well as the subsequent response following the lunch meal.

DETAILED DESCRIPTION:
Twelve habitual breakfast consumers with type 2 diabetes (T2D) were recruited for the study. They completed two, 7-day conditions in random order with a minimum of a 7-day washout period between study days. They consumed either a high protein (PRO) or high carbohydrate (CHO) breakfast for 6 days of acclimatization, and on the seventh day, they reported to the lab at 0700 hours following a ~12 hour overnight fast and underwent forearm catheterization before a baseline blood draw. The participants consumed the respective breakfast at ~0730 hours. Four hours post-breakfast, subjects consumed a standard lunch meal. Blood samples were taken continuously throughout the 8-hour test day.

ELIGIBILITY:
Inclusion Criteria:

* 21-55 y of age
* body mass index (BMI) between 30-40 kg/m2
* weight stable for the prior 6 months
* non-smokers
* minimal alcohol consumption (< 2 drinks per day)
* type 2 diabetic (diagnosed ≥ 2 y)
* a fasting glucose level above 120 mg/dL
* HbA1c between 6.5-9.0%

Exclusion Criteria:

* insulin
* β-blockers
* GLP-1 agonists (e.g. exenatide)
* dipeptidyl peptidase (DPP) inhibitors
* weight loss
* using weight-loss medications
* pregnant or lactating

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park YM, Heden TD, Liu Y, Nyhoff LM, Thyfault JP, Leidy HJ, Kanaley JA. A high-protein breakfast induces greater insulin and glucose-dependent insulinotropic peptide responses to a subsequent lunch meal in individuals with type 2 diabetes. J Nutr. 2015 Mar;145(3):452-8. doi: 10.3945/jn.114.202549. Epub 2014 Dec 24. PMID 25733459

RESULTS

PARTICIPANT FLOW:
Groups:
- High Carb Then High Protein Breakfast: A high carbohydrate breakfast for 7 days, followed by a 7-day washout, followed a high protein breakfast for 7 days
- High Protein Then High Carb Breakfast: A high protein breakfast for 7 days, followed by a 7-day washout, followed a high carbohydrate breakfast for 7 days
Period: First Intervention (7 Days)
Arm/Group | High Carb Then High Protein Breakfast | High Protein Then High Carb Breakfast
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Washout (7 Days)
Arm/Group | High Carb Then High Protein Breakfast | High Protein Then High Carb Breakfast
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Second Intervention (7 Days)
Arm/Group | High Carb Then High Protein Breakfast | High Protein Then High Carb Breakfast
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- High Carb Then High Protein Breakfast: A high carbohydrate breakfast - 500 kcal (15% protein, 65% CHO, 20% fat) for 7 days, followed by 7-day washout, followed by a high protein breakfast for 7 days
- High Protein Then High Carb Breakfast: A high protein breakfast - 500 kcal (35% protein, 45% CHO, 20% fat) for 7 days, followed by a 7-day washout, followed by a high carbohydrate breakfast for 7 days
- Total: Total of all reporting groups
Arm/Group | High Carb Then High Protein Breakfast | High Protein Then High Carb Breakfast | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Plasma Glucose Level Post-meal (AUC [0-4])
Description: AUC for 4 hr after breakfast and after lunch
Time Frame: 0-240 and 240-480
Measure: Mean (Standard Error); unit: min*pg/ml
Groups:
- High Protein Breakfast: a high protein breakfast - 500 kcal (35% protein, 45% CHO, 20% fat)
  high protein breakfast
  high carbohydrate breakfast
- High Carbohydrate Breakfast: a high carbohydrate breakfast - 500 kcal (15% protein, 65% CHO, 20% fat)
  high protein breakfast
  high carbohydrate breakfast
Arm/Group | High Protein Breakfast | High Carbohydrate Breakfast
Number analyzed (Participants) | 12 | 12
min*pg/ml | 28426 (1660) | 33911 (2590)

2. Secondary Outcome: Post-meal Level of Glucose-dependent Insulinotropic Peptide (GIP) (AUC)
Description: AUC for 4 hr after breakfast and after lunch
Time Frame: 0-240 and 240-480
Measure: Mean (Standard Error); unit: min*pg/ml
Arm/Group | High Protein Breakfast | High Carbohydrate Breakfast
Number analyzed (Participants) | 12 | 12
min*pg/ml | 15156 (3100) | 14620 (1814)

3. Other Pre Specified Outcome: Post-meal Insulin Level (AUC [0-4])
Description: AUC for 4 hr after breakfast and after lunch
Time Frame: 0-240 and 240-480
Measure: Mean (Standard Error); unit: min*pg/ml
Arm/Group | High Protein Breakfast | High Carbohydrate Breakfast
Number analyzed (Participants) | 12 | 12
min*pg/ml | 428869 (55831) | 474236 (53518)

4. Other Pre Specified Outcome: Post-meal Glucagon-like Peptide-1 (GLP-1) Level (AUC )
Description: AUC for 4 hr after breakfast and after lunch
Time Frame: 0-240 and 240-480
Measure: Mean (Standard Error); unit: ng/ml x min for 4 h
Arm/Group | High Carb Then High Protein Breakfast | High Protein Then High Carb Breakfast
Number analyzed (Participants) | 12 | 12
ng/ml x min for 4 h | 14 (3.1) | 11.5 (2)

ADVERSE EVENTS:
Arm/Group | High Protein Breakfast | High Carbohydrate Breakfast
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No